CLINICAL TRIAL: NCT02907125
Title: Strengthening the Evidence Base on Effective scHool Based intErventions for pRomoting Adolescent Health (SEHER)
Brief Title: Extended Evaluation of School-based Health Promotion Programmes in Bihar, India
Acronym: SEHER+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sangath (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); Public Health Foundation of India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SANSEHER2016_0001
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Last update posted 2020-12-10 (Actual); Status verified 2017-05

CONDITIONS: Health Promotion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TSM arm (Experimental): The SEHER intervention will be delivered by a trained teacher, called as Teacher-as-SEHER Mitra (Mitra meaning friend) or lay health worker called as SEHER Mitra being trained to facilitate following activitiesAwareness generation activities for all stakeholders in school; Wall-magazine, Speak-out box, Competitions, School Health Promotion Committee, School health policies, Peer groups of students of class IX and X students, Workshops and talks for all the students from standard IX, and for teachers, and Counselling and referral services for all the students in the school.
  This intervention will be delivered in each school over the academic year.
  Interventions: Behavioral: SEHER Intervention delivered by TSM; Behavioral: Tarang AEP
- SM arm (Experimental): The SEHER intervention will be delivered by a lay health worker called as SEHER Mitra being trained to facilitate following activities: Awareness generation activities for all stakeholders in school; Wall-magazine, Speak-out box, Competitions, School Health Promotion Committee, School health policies, Peer groups of students of class IX and X students, Workshops and talks for all the students from standard IX, and for teachers, and Counselling and referral services for all the students in the school.
  This intervention will be delivered in each school over the academic year.
  Interventions: Behavioral: SEHER Intervention delivered by SM; Behavioral: Tarang AEP
- Comparison arm Tarang AEP (Active Comparator): The comparison arm involves 'usual care' which in the study setting is the Tarang: Adolescence Education Programme comprising of 16 classroom sessions on process of growing-up, prevention of HIV/AIDS and other Sexually Transmitted Diseases (STDs), and prevention of substance and other drug abuse. This programme is delivered by a trained nodal teacher in the school over the academic year.
  Interventions: Behavioral: Tarang AEP

INTERVENTIONS:
Behavioral: SEHER Intervention delivered by TSM — SEHER Intervention The SEHER intervention will be delivered by a trained teacher, called as Teacher-as-SEHER Mitra (Mitra meaning friend) or lay health worker called as SEHER Mitra being trained to facilitate following activitiesAwareness generation activities for all stakeholders in school; Wall-magazine, Speak-out box, Competitions, School Health Promotion Committee, School health policies, Peer groups of students of class IX and X students, Workshops and talks for all the students from standard IX, and for teachers, and Counselling and referral services for all the students in the school.
  This intervention will be delivered in each school over the academic year.
  Other Names: TSM Arm
  Arms: TSM arm
Behavioral: SEHER Intervention delivered by SM — The SEHER intervention will be delivered by a lay health worker called as SEHER Mitra being trained to facilitate following activities: Awareness generation activities for all stakeholders in school; Wall-magazine, Speak-out box, Competitions, School Health Promotion Committee, School health policies, Peer groups of students of class IX and X students, Workshops and talks for all the students from standard IX, and for teachers, and Counselling and referral services for all the students in the school.
  This intervention will be delivered in each school over the academic year.
  Other Names: SM arm
  Arms: SM arm
Behavioral: Tarang AEP — The comparison arm involves 'usual care' which in the study setting is the Tarang: Adolescence Education Programme comprising of 16 classroom sessions on process of growing-up, prevention of HIV/AIDS and other Sexually Transmitted Diseases (STDs), and prevention of substance and other drug abuse. This programme is delivered by a trained nodal teacher in the school over the academic year.
  Other Names: Comparison arm

SUMMARY:
SEHER Plus- Strengthening Evidence base on scHool-based intErventions for pRomoting adolescent health, seeks to evaluate a school based adolescent health promotion intervention delivered by two different delivery agents viz. teacher-as-SEHER Mitra (TSM) and lay school counsellor called as SEHER Mitra (SM) in government- run secondary schools in Bihar, India. SEHER Plus will be implemented in the same randomly assigned 74 schools wherein, the SEHER trial (ClinicalTrials.gov ID: NCT02484014)-a three armed clustered randomised trial (CRT) was implemented to evaluate the effectiveness and cost-effectiveness of these two models compared with the Tarang-Adolescence Education Programme (usual care) implemented by the State Government of Bihar.

The SEHER trial hypothesised that both interventions, compared to the control arm, would lead to a greater impact on school climate (school connectedness and relationship with teachers and fellow students). In addition, the interventions would increase the knowledge, attitude and awareness, and promoting healthy behaviours in youth on reproductive and sexual health outcomes, mental health and substance use, and gender related attitudes and violence. The SEHER trial also hypothesized that the addition of more resource intensive component (the SM arm) would be associated with the best outcomes. The hypothesis for the SEHER Plus is that students who will have exposure to the SEHER intervention activities in two academic years (Class IX and X) will show greater benefits on the primary, secondary and exploratory outcomes than students who have exposure to the SEHER intervention activities in one academic year (Class IX).

DETAILED DESCRIPTION:
Background and objective: India is home to 358 million young people in the age group of 10 to 24; of these 243 million are between 10 and 19 years age. This represents a huge opportunity that can transform the social and economic fortunes of the country. Key public health challenges for adolescents in India include unwanted pregnancies, sexually transmitted and reproductive tract infections, injuries, growing misuse of alcohol, tobacco and other substances, and mental health problems such as depression, anxiety disorders and suicide. Schools provide an ideal platform for addressing these health issues and the World Health Organization's Health Promoting Schools framework seeks to address some of the structural determinants of these health concerns. The recent Cochrane review assessed school- based interventions and found that 'whole school' or 'school environment' interventions are effective in addressing a range of health outcomes among adolescents including bullying, aggression, and tobacco use. However, there is no comparable evidence on effectiveness and cost-effectiveness on school-based health promotion programmes in India.

Sangath has implemented SEHER-Strengthening Evidence base on school-based intErventions for pRomoting adolescent health (ClinicalTrials.gov ID: NCT02484014) , which is a jointly funded programme (by The MacArthur Foundation and United Nation's Population Development Fund, India) that seeks to develop and evaluate a comprehensive adolescent health promotion intervention delivered by two different delivery agents viz. teacher as SEHER Mitra (TSM) and a lay health worker called as SEHER Mitra (SM) in government run secondary schools in Bihar, India. Following hypotheses are addressed through SEHER trial:

1. For primary outcome measure: It is hypothesized that the intervention strategies in addition to usual intervention (Tarang-AEP) will have a graded effect on overall school climate.
2. For secondary outcome measures: The interventions will build positive attitude towards gender equity, build knowledge of and attitude towards reproductive and sexual health, reduce self-reported bullying, violence and depression.
3. For exploratory outcome measures : The interventions will decrease tobacco, alcohol and other substance use, reduce suicide behaviour (suicide thoughts and attempts) and increase safe sexual behaviour.

Hypotheses for SEHER Plus:

The SEHER Plus will address the additional benefits of providing an exposure to intervention activities for two years versus one year.

For primary outcome measure: The students who will have exposure to the SEHER intervention activities in addition to the usual intervention (Tarang-AEP) in two academic years (Class IX and X) will show greater benefits on overall school climate than students who have exposure to the SEHER intervention activities and usual intervention (Tarang-AEP) in one academic year (Class IX).

For secondary outcome measures: The students who will have exposure to the SEHER intervention activities in addition to the usual intervention (Tarang-AEP) in two academic years (Class IX and X) will show improved positive attitude towards gender equity, increased knowledge of and attitude towards reproductive and sexual health, reduced self-reported bullying, violence and depression than students who have exposure to the SEHER intervention activities and usual intervention (Tarang-AEP) in one academic year (Class IX).

For secondary outcome measures: The students who will have exposure to the SEHER intervention activities in addition to the usual intervention (Tarang-AEP) in two academic years (Class IX and X) will report reduced incidence of tobacco, alcohol and other substance use, reduced incidence of self-reported suicide attempts and reduced incidence of sexual behaviour than students who have exposure to the SEHER intervention activities and usual intervention (Tarang-AEP) in one academic year (Class IX).

The SEHER intervention with the already existing Tarang-AEP will enhance the effect on the above mentioned outcomes; the effects will be minimal to moderate among the students who have two years exposure and are from low resource intensity intervention (Teacher-as-SEHER Mitra: Arm-I), and the effects will be the greatest and significant among the students who have two years exposure and are from high resource intensity intervention (School Mitra: Arm-II).

Randomisation: The school as the unit of randomisation are allocated to one of the intervention arms or comparison using minimisation during the pilot study of the SEHER project (June 2014-March 2015). Although, usually a pilot study would be conducted in different schools from those in the main trial, it has been possible for SEHER to conduct the pilot study in the main trial schools because a new cohort of standard IX students will be entering school every year.

Before randomisation, a list of eligible schools for randomisation (n=112) from the total number of secondary and higher secondary schools in Nalanda district of Bihar (n=136) was generated. The following criteria were used to generate the list: implementation of Tarang-AEP programme, total number of students in the school, and total number of employed teachers in school.

Of the 112 schools, 75 were randomly selected for the random allocation. To have a representative pool of 75 schools, and to ensure an equal number of schools of each type in each of the three trial arms, 68 % of co-educational (63 out of 93), 69% of only girls' (9 out of 13) and 50% only boys' schools (3 out of 6) were selected. All the 75 schools are allocated to comparison or one of the intervention arms by using minimization. To carry out the allocation by minimisation, the arms were balanced on the following variables (each of the variable will be classified into categories):

1. Type of school (secondary= 1; and secondary and higher secondary school= 2);
2. School size (small=100-300; medium=301-600, and large=601 and above students ), and
3. Nature of school (Co-education=1; only boys'=2; and only girls' =3). The random allocation by using minimization was carried out by an independent statistician (Gian Luca DiTanna, LSHTM) using the R software package .

One school from the TSM arm dropped out after the pilot study and hence there are now 24 schools in this arm.

Sample size: All the students who are enrolled in class IX in the academic year March 2015- April 2016 and all the students who are enrolled in the class IX in the academic year March 2016- April 2017 will be invited to participate in the outcome assessment to be completed in December 2016/January 2017.

The investigators will not collect any baseline assessment for the students who are enrolled in Class IX in the academic year 2016-17. As part of the SEHER trial, the students who are enrolled in class IX in the academic year 2015-16 have participated in two outcome assessments; one in July 2015 and other in March/April 2016.

Process Evaluation: Process evaluation will be an integral part of the research design and will examine the quality of programme implementation (i.e. its integrity or fidelity), the completeness of its delivery, and the extent to which stakeholders engage with it. In doing so, it can help explain the programme's outcomes and identify ways to improve and/or replicate it. Two types of indicators will be collated to evaluate the fidelity of the delivery of the SEHER interventions, viz. their quantity and quality.

Nested qualitative evaluation: A qualitative evaluation will be conducted at the end of the intervention to: a) explore deliverers' and recipients' responses to the intervention, and b) explore the school communities perception about the effect of the SEHER intervention on the students' health and academic attainment. The qualitative component will comprise of focus group discussions with single sex groups of class IX and X students, TSMs and SMs, and in-depth interviews with purposively selected male and female students from class IX and X who have availed counselling services, principals, Tarang nodal teachers and other teachers, TSMs/SMs and supervisors.

Data management: Two types of quantitative data will be collected: intervention process, and outcome assessment. All outcome assessment data will be collected in paper form, as will process data from TSMs/SMs. All the data will be manually entered into Access database. Range and consistency checks will be performed at monthly intervals for all process data. Queries identified will be resolved promptly by the trial management team, and the database updated, maintaining the audit trail. All data will be kept in separate databases and only merged into a master database after data collection is completed and each individual database will be locked. All process data will be backed-up on external hard disks on monthly basis. Access to pre-locked data will be password protected at multiple levels and no member of the trial team apart from the data manager and independent statistician will have access to these passwords. After the dataset is locked, the dataset will remain password-protected and trial investigators will have access to the datasets. For all data, a separate file linking names and trial identification codes will be kept and password protected.

Analysis:Quantitative analyses will be carried out using STATA (version 14). Below is a summary of the investigator's approach to the analysis. A detailed analysis plan will be agreed with the Data Safety and Monitoring Board towards the end of the trial and/or before any analysis is undertaken.

Descriptive analyses: Initial analyses will describe the characteristics of enrolled participants within and across arms (for example: age and socioeconomic background).

The outcome measures will be summarised at end-line by each cluster, arm-wise and year-wise exposure, and overall. These will be summarised by means (SD), medians (Inter- Quartile Range) or numbers and proportions as appropriate by key relevant subgroups (such as age, and gender).

Outcome analyses: The primary analyses, based on cross sectional survey, will be intention-to-treat at the end of the trial and using multi-level modelling to take into account clustering at the school level. Gender-wise sub-group analysis will be performed. The trial outcomes will be evaluated for the primary and secondary outcomes based on the change in the intervention arm compared to the change in the comparison. The primary trial impact comparison will be arm-wise analysed between the the students who have exposure to intervention activities for two academic years and the students who have exposure to intervention activities for one academic year.

Mixed effects regression will be performed to analyse changes in primary and secondary outcomes at school-level. Effect sizes will be presented as risk ratios for binary outcomes (for e.g. experience of bullying), and as mean differences for continuous outcomes (for e.g. overall school climate score); 95% confidence intervals (CI) will be derived for both.

The reporting and presentation of this trial will be in accordance with the CONSORT guidelines for cluster randomised trials, with the primary comparative analysis being conducted on an intention-to-treat basis.

ELIGIBILITY:
Inclusion Criteria:

* All the students enrolled in class IX in academic year March 2015- April 2016 and enrolled in class IX in academic year March 2016- April 2017 in all the randomly assigned 74 schools will be invited to participate in the study.

Exclusion Criteria:

* None

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29527 (Actual)
Dates: Start 2016-06-15; Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
School Climate | Up to 7 months
  The school climate will be measured through Beyond Blue School Climate Scale (28 items)

SECONDARY OUTCOMES:
Self-reported bully behaviour | Up to 7 months
  The bully behaviour will be measured through adapted version of Illinois Bullying Scale (4 items)
self-reported violence | Up to 7 months
  This outcome measure will be assessed through adapted version of Global School-based student Health Survey (4 items)
Attitude towards gender equity | Up to 7 months
  This outcome measure will be assessed through adapted version of Gender Equitable Men Survey (GEMS) 10 items.
Knowledge and attitude towards Reproductive and Sexual Health | Up to 7 months
  This outcome measure will be assessed through 10 self-reported items based on the WHO's illustrative questionnaire for interview/survey with young people
Depression | Up to 7 months
  This outcome will be assessed through the Patient Health Questionnaire-9

OTHER OUTCOMES:
Self-reported substance use | Up to 7 months
  This outcome will be assessed through adapted version of Global School-based student Health Survey
Self-reported sexual behaviour | Up to 7 months
  This outcome will be assessed through adapted version of Global School-based student Health Survey
Self-reported suicide attempts | Up to 7 months
  This outcome will be assessed through adapted version of Global School-based student Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Patel, FMedSci, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Sangath, Bardez, Goa, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shinde S, Weiss HA, Khandeparkar P, Pereira B, Sharma A, Gupta R, Ross DA, Patton G, Patel V. A multicomponent secondary school health promotion intervention and adolescent health: An extension of the SEHER cluster randomised controlled trial in Bihar, India. PLoS Med. 2020 Feb 11;17(2):e1003021. doi: 10.1371/journal.pmed.1003021. eCollection 2020 Feb. PMID 32045409